CLINICAL TRIAL: NCT01732198
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Immunogenicity, Reactogenicity, and Safety Study of NU300 Booster Dose Compared to ActHIB®, Both Co-administered With Prevnar 13® at 12-15 Months of Age, in Healthy Toddlers Who Have Received a Primary Series of a Licensed Hib Vaccine and Prevnar 13®
Brief Title: A Phase 2, Multicenter, Open-label Study to Assess the Immunogenicity of an Investigational Hib Vaccine (NU300)in Toddlers
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nuron Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CP-NU300-02
Record Dates: First submitted 2012-11-19; First posted 2012-11-22 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Infectious Disease
MeSH Terms: conditions — Communicable Diseases | interventions — Haemophilus influenza type b polysaccharide vaccine-tetanus toxin conjugate; 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NU300 and Prevnar 13 (Experimental): NU300 at a single dose of 0.5 mL IM
  Interventions: Biological: NU300; Biological: Prevnar 13
- ActHIB and Prevnar 13 (Active Comparator): ActHIB at a dose of 0.5 ml IM
  Interventions: Biological: ActHIB; Biological: Prevnar 13

INTERVENTIONS:
Biological: NU300
  Arms: NU300 and Prevnar 13
Biological: ActHIB
  Arms: ActHIB and Prevnar 13
Biological: Prevnar 13

SUMMARY:
Evaluate the safety and tolerability of a single booster dose of NU300, co-administered with Prevnar 13® over a 28 day period following the injection compared to a single booster of ACTHIB co-administered with Prevnar 13® over a 28 day period following the injection.

Evaluate the immunogenicity, as determined by anti-PRP polysaccharide response, of a single booster dose of NU300 co-administered with Prevnar 13® compared to a single booster dose of ActHIB® co-administered with Prevnar 13®.

Evaluate the individual IgG antibody quantitative response to the 13 antigens in Prevnar 13® following NU300 co-administration with Prevnar 13® compared to the IgG antibody response to the pneumococcal polysaccharides following ActHIB® co-administration with Prevnar 13® 28 days following injection.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained from the parent or guardian of the subject
2. Male or female subjects 12-15 months of age at the time of booster vaccination, who had previously received complete primary vaccination series with a licensed Hib product and Prevnar 13® in accordance with the FDA approved labels.
3. Subjects for whom the investigator believes that the parent/guardian can and will comply with the requirements of the protocol
4. Subjects free of obvious health problems as established by medical history and clinical examination before entering the study

Exclusion Criteria:

1. Previous booster vaccination against Hib and/or Prevnar 13®
2. Any confirmed or suspected Haemophilus influenzae or pneumococcal illness.
3. Administration of a vaccine not foreseen by the study protocol during the period starting from 30 days before and ending 28 days after administration of study vaccines (before the blood draw at Visit 2).
4. Chronic administration of immunosuppressants or other immune-modifying drugs within 30 days prior to dosing in the study.
5. Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and/or clinical examination.
6. Early pre-term birth (delivery before 32 weeks).
7. Major congenital defects or serious chronic diseases, or serious conditions including history of seizures, apnea, etc.
8. Concurrent participation in another clinical study at any time during the study period or within the previous 6 months in which the subject has been or will be exposed to an investigational or non-investigational product (pharmaceutical product, formula, or device)
9. Presence of a moderate or severe illness with or without fever at the time of vaccination (fever is defined as a temperature of ≥ 38.0C [100.4F]).
10. Known history of thrombocytopenia or any coagulation disorder.
11. Known hypersensitivity to any of the components of the vaccines.
12. Known hypersensitivity to latex.
13. The subject is unable to provide an adequate blood draw for immunogenicity assays, and safety panels at Visit 1

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-01 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
safety and efficacy | one month
  Evaluate the safety and tolerability of a single booster dose of NU300, co-administered with Prevnar 13® compared to a single booster dose of ActHIB® co-administered with Prevnar 13®, over a 28 day period following injection
  Evaluate the immunogenicity, as determined by anti-PRP polysaccharide response, of a single booster dose of NU300 co-administered with Prevnar 13® compared to a single booster dose of ActHIB® co-administered with Prevnar 13®.

SECONDARY OUTCOMES:
Evaluate the individual IgG antibody quantitative response to the 13 antigens in Prevnar 13® | one month
  Evaluate the individual IgG antibody quantitative response to the 13 antigens in Prevnar 13® following NU300 co-administration with Prevnar 13® compared to the IgG antibody response to the pneumococcal polysaccharides following ActHIB® co-administration with Prevnar 13® 28 days following injection

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Oakland, California
  - Bardstown, Kentucky